CLINICAL TRIAL: NCT04698616
Title: The Relation Between Lean Body Mass and Side Effects Induced by Chemotherapy in Patients With Lymphoma: A Prospective Cohort Study
Brief Title: Lean Body Mass and Side Effects in Patients With Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Sponsor - Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: SJ-823
Record Dates: First submitted 2020-05-28; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Malignant Lymphoma
Keywords: lymphoma; body composition; lean body mass; chemotherapy; quality of life (QOL); nutritional status; physical activity
MeSH Terms: conditions — Lymphoma; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malignant lymphoma patients: Identification of the patients who are/are not dose-reduced due to chemotherapy, and then look at the body composition in connection with this.

SUMMARY:
The primary purpose is to investigate the relationship between the dose of chemotherapeutic agents per kilogram of lean body mass (LBM) and the development of side effects induced by chemotherapy in patients with lymphoma. Secondarily, the maximum tolerable dose of chemotherapeutics (MTD), patients' quality of life (QOL), nutritional status and physical activity during the course of treatment are estimated.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving myelosuppressive treatment for malignant lymphoma assessed by the investigator.
* Legal of age

Exclusion Criteria:

* ECOG Performance Status ≥2
* People who cannot speak and understand Danish
* Pregnant and breastfeeding
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving myelosuppressive treatment for malignant lymphoma
Sampling Method: Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-03-03 (Estimated)

PRIMARY OUTCOMES:
Lean Body Mass (LBM) | 8 weeks (two treatment cycles)
  LBM measured by bioelectrical impedans corelated to the dosis of chemotherapeutics given

SECONDARY OUTCOMES:
Maximal tolerable dose of chemotherapeutics (microg/ml/kg LBM), | 8 weeks (two treatment cycles)
  Patients with side effects - correlation between dose of cytostatics/ kg LBM compared to patients without side effects
Quality of life (QOL) (score EORTC) | 8 weeks (two treatment cycles)
  Correlation of score and difference in LBM (kg)
nutritional status at inclusion (NRS2002 - scale) | 8 weeks (two treatment cycles)
  Predictive value of scale for ocurrence of side-effects (binary)
physical activity (scale - questionaire) | 8 weeks (two treatmenr cycles)
  Corelation between cytostatic dose/kg LBM and scale

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD,MPA, Study Chair — University of Copenhagen
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen, Frederiksberg
  - Sjællands Universitetshospital, Hæmatologisk Afdeling H60, Roskilde

IPD SHARING:
Plan to Share IPD: No